CLINICAL TRIAL: NCT06904755
Title: Clinical Study on Safety and Effectiveness of Mesenchymal Stem Cells in Blood Purification for the Treatment of Liver Failure
Brief Title: Safety and Effectiveness of Mesenchymal Stem Cells in Blood Purification for the Treatment of Liver Failure
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kebo Zhong (Other)
Responsible Party: Sponsor-Investigator, Kebo Zhong, doctor, Zhujiang Hospital
Organization: Zhujiang Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhujiang Hospital
Record Dates: First submitted 2025-01-07; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood purification with mesenchymal stem cells therapy group (Experimental)
  Interventions: Device: It is loaded with a mesenchymal stem cells reaction device for blood purification

INTERVENTIONS:
Device: It is loaded with a mesenchymal stem cells reaction device for blood purification — Artificial liver blood purification therapy is performed using a mesenchymal stem cells reactor.

SUMMARY:
The goal of this clinical trial is to learn if mesenchymal stem cells in blood purification works to treat liver failure in adults. It will also learn about the safety and effectiveness of mesenchymal stem cells in blood purification. The main questions it aims to answer are:1.Does mesenchymal stem cells in blood purification improve the condition of patients with liver failure? 2.What medical problems do participants have when taking mesenchymal stem cells in blood purification? Participants will receive routine medical treatment and blood purification treatment with mesenchymal stem cells.These cells work outside the body and do not enter the body. We will: 1.Collect samples from participants such as blood, Urine and feces. 2.record post-treatment outcomes such as survival rate at 4 weeks after treatment, conversion rate to liver transplantation, Inflammatory, survival rate at 7days, 14days, 8 weeks and 12 weeks after treatment, and liver disease indicators(prothrombin time activity percentage, lactic aicd, blood ammonia, α-fetoprotein, ferritin).

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 65 years old;
2. Patients with acute liver failure in the early and intermediate stages caused by various reasons;
3. Total bilirubin (TBil) ≥ 171μmol/L or an increase of ≥ 17.1μmol/L per day;
4. Prothrombin activity (PTA) between 20% and 40% (or INR between 1.5 and 2.6);
5. No hepatic encephalopathy or encephalopathy below grade II (including grade II);
6. Elevated inflammatory markers (IL-6 / TNF-α / CRP, etc.);
7. The subjects are able to communicate well with the researchers and can complete the study in accordance with the study regulations;
8. The subjects must be informed of this study and voluntarily sign a written informed consent form before the experiment.

Exclusion Criteria:

1. Patients with severe active bleeding or diffuse intravascular coagulation;
2. Patients with a high degree of allergy to blood products or drugs used during treatment, such as plasma, heparin, and protamine;
3. Patients with circulatory failure;
4. Patients with a MELD score > 30;
5. Patients with other severe heart diseases, lung diseases, blood diseases, autoimmune diseases, or diabetes;
6. Subjects who may be unable to complete this study for other reasons or who the researchers believe should not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival rate on day 28 after treatment | From enrollment to day 28 after treatment.
  researchers record all participators' survival condition from enrollment to day 28 after treatment.

SECONDARY OUTCOMES:
conversion rate to liver transplantation | From enrollment to day 28, 56, 84 after treatment.
  researchers record participators' condition of conversion to liver transplantation from enrollment to day 28, 56, 84 after treatment.
Interleukin-6(IL-6) | From enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
  Participators accept blood tests of a Inflammatory factor: reflect systemic inflammatory status.
Survival rate on day 7, 14, 56, 84 after treatment | From enrollment to day 7, 14, 56, 84 after treatment.
  Researchers record participators' survival condition from enrollment to day 7, 14, 56, 84 after treatment.
lactic aicd | From enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
  Participators accept blood tests of liver disease indicators lactic aicd from enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
Model for End-Stage Liver Disease score | From enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
  The internationally recognized prognostic scoring system for end-stage liver disease is used to determine prioritization for liver transplantation and predict patient survival rates.
Chinese group on the study of severe hepatitis B-acute-on-chronic liver failure score | From enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
  To assess short-term mortality rates (28-day/90-day) in patients with acute-on-chronic liver failure (ACLF) and guide prioritization for liver transplantation and intensive care resource allocation.
tumor necrosis factor α (TNF-α) | From enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
  Participators accept blood tests of a Inflammatory factor: reflect systemic inflammatory status.
C-reactive protein (CRP) | From enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
  Participators accept blood tests of a Inflammatory factor: reflect systemic inflammatory status.
blood ammonia | From enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
  Participators accept blood tests of liver disease indicators blood ammonia from enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
Alpha-fetoprotein (AFP) | From enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
  Participators accept blood tests of liver disease indicators AFP from enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
ferritin | From enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
  Participators accept blood tests of liver disease indicators ferritin from enrollment to day 1, 3, 5, 7, 14, 28, 56, 84 after treatment.
Incidence rate of adverse events (AE incidence rate) | Throughout the entire course of MSC-based blood purification therapy.
  Record treatment-related adverse reactions occurring during the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
We fully acknowledge the significance of data sharing. However, owing to the policies and confidentiality agreements adhered to in our laboratory, we regretfully cannot furnish the raw data. Nevertheless, we have meticulously presented a comprehensive account of the experimental design, analysis, results, and the procedures employed for data analysis and processing.